CLINICAL TRIAL: NCT07229573
Title: The Effectiveness of Serious Game-Based Training for Nursing Students in Postpartum Haemorrhage Management: A Randomised Controlled Trial
Brief Title: The Effectiveness of Serious Game-Based Training for Nursing Students in Postpartum Haemorrhage Management
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sakarya University (Other)
Responsible Party: Principal Investigator, Ahsen Demirhan, PhD, Sakarya University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 06.10.2025
Record Dates: First submitted 2025-11-13; First posted 2025-11-17 (Actual); Last update posted 2025-11-17 (Actual); Status verified 2025-11

CONDITIONS: Gamification; Gamification in Health Education; Nurse Education; Nursing Students; Postpartum Hemorrhage; Nursing Care
MeSH Terms: conditions — Postpartum Hemorrhage

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Gamification Group (Experimental): Students in the intervention group will first receive traditional theoretical and practical training in the department's curriculum using standard methods; they will then participate in the developed serious game application.
  Interventions: Other: Gamification
- Control Group (No Intervention): Students in the control group will only receive theoretical and practical lessons included in the department curriculum using traditional teaching methods during the study period; no additional intervention will be applied. The scope of education will be limited to the existing course content, and no additional simulation/game-based activities will be conducted. In accordance with ethical principles, the same serious game application will be offered to the students in the control group after the research is completed, and these students will also be provided with the opportunity to benefit from the game.

INTERVENTIONS:
Other: Gamification — Students in the intervention group will first receive traditional theoretical and practical training in the department's curriculum using standard methods; they will then participate in the developed serious game application.
  Arms: Gamification Group

SUMMARY:
This randomised controlled trial aims to evaluate the effectiveness of serious game-based training for postpartum haemorrhage (PPH) management among third-year nursing students. The study employs a pre-test-post-test design with two parallel groups: an experimental group (game-based education) and a control group (traditional education). The sample size was determined by power analysis to be 70 students in total, with 35 students in each group. Participants will be assigned in a 1:1 ratio by computer-assisted block randomisation by a person independent of the research team; students and instructors will not be blinded, but the biostatistician performing the data analysis will be blinded. The intervention group will first receive traditional education, followed by gamification-based education including nursing interventions in the management of PPB; the control group will receive only traditional education. Data will be collected using the PPK Management Knowledge and Skills Assessment Form and the PPK Management Self-Confidence Scale.

ELIGIBILITY:
Inclusion Criteria:

a) Third-year nursing students taking the Obstetrics and Gynaecology Nursing course, b) Not experiencing any verbal or written communication problems, c) Not being an exchange student, d) Being willing to provide written consent before participating in the study.

Exclusion Criteria:

Not meeting the inclusion criteria

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2025-11-05 (Actual); Primary Completion 2025-11-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Postpartum Haemorrhage Management Knowledge and Skills | pre-education and within 1 week after training
  The form was developed by researchers for this study based on the literature. The assessment form, consisting of 20 multiple-choice questions, was prepared to evaluate the student's knowledge and skill levels in PPB management. The opinions of three experts in the field of Women's Health and Obstetric Nursing and Midwifery were sought to assess the comprehensiveness, clarity, and scientific appropriateness of the questions on the form. In the Postpartum Haemorrhage Management Knowledge and Skills Assessment Form, each correct answer is scored as '5' and each incorrect answer as '0'. The maximum score that can be obtained from the form is "100", and the minimum score is '0'.
Self-Confidence Scale in PPH Management | pre-education and within 1 week after training
  The form was developed by researchers for this study based on the literature. The assessment form, consisting of 10 multiple-choice questions, was prepared to evaluate the student's level of self-efficacy in PPH management.
  Three experts in the field of Women's Health and Obstetric Nursing and Midwifery were consulted to assess the comprehensiveness, clarity, and scientific appropriateness of the questions on the form. The scale is a 5-point Likert scale (1=Strongly disagree 2=Disagree 3=Undecided 4=Agree 5=Strongly agree)
Self-Regulated Learning Scale for Clinical Nursing Practice | pre-education and within 1 week after training
  The scale was developed by Satoko Iyama and Hitomi Maeda in 2017 and adapted into Turkish by Şenol and Orgun in 2018. It consists of 16 items in a 5-point Likert scale type, comprising two sub-dimensions: 'Motivation' and 'Learning Strategies'. The scale is structured as follows: 1. Motivation 2. Learning Strategies It is a 5-point Likert-type scale comprising 16 items and two subscales: 'Motivation' and "Learning Strategies". The minimum score achievable on the entire scale is 16, with a maximum score of 80, and Cronbach's α was determined to be 0.898.

CONTACTS AND LOCATIONS:
Locations (1):
- Sakarya University, Adapazarı, Sakarya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No